CLINICAL TRIAL: NCT07388654
Title: Adapting a Brief Dyadic Intervention for Co-occurring Post-Traumatic Stress Disorder and Alcohol Use Disorder
Brief Title: PTSD and Alcohol Couples Treatment for Veterans
Acronym: PACT-V
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRD9-003-24W; IK2RD000536 (Other Grant/Funding Number: RRDT)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: PTSD, AUD
Keywords: Stress Disorders, Post-Traumatic; Alcohol Use Disorder; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Intervention Model Description: This is a stage 1a/1b one-armed non-randomized pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COPE + BFIT (Experimental): In this single arm study, participants will be assigned only to the pilot intervention of COPE + B-FIT.
  Interventions: Behavioral: COPE + BFIT

INTERVENTIONS:
Behavioral: COPE + BFIT — Veterans will engage in 12 sessions of COPE individually, and Veterans and their significant others will participate in in 3-4 sessions of the adapted B-FIT intervention specifically for Veterans with PTSD + AUD and their partners. COPE will be delivered concurrently with the adapted B-FIT.
  Other Names: Concurrent Treatment of PTSD and Substance Use Disorder with Prolonged Exposure and Brief Family Involved Treatment

SUMMARY:
Treatment of post-traumatic stress disorder (PTSD) and alcohol use disorder (AUD) treatment for Veterans is challenging for Veterans. Veterans often benefit from social support from friends and loved ones while in treatment; however, the symptoms of PTSD and AUD often are associated with increased relationship conflict. It is essential to identify new ways to improve PTSD-AUD treatment, and involving loved ones in the process may be a way to improve treatment.

The purpose of this study is to pilot test a brief couples intervention that is designed to be delivered while Veterans are in treatment for PTSD-AUD. Over the course of 12 weeks, Veterans will receive individual treatment through Concurrent Treatment of PTSD and Substance Use Disorders with Prolonged Exposure (COPE), and Veterans and their romantic partners will attend 3-4 sessions of Brief Family Involved Treatment (B-FIT) which has been modified specifically for Veterans with PTSD-AUD. Veterans and their romantic partners will complete a baseline visit, 12 weeks of weekly measures, and a 3-month follow-up visit. This is a stage 1a one-armed non-randomized pilot trial.

DETAILED DESCRIPTION:
Co-occurring PTSD-AUD is a complex and urgent public health crisis. COPE is a highly efficacious integrated intervention that has strong positive effects on reducing PTSD symptoms, but has substantial room for improvement regarding AUD outcomes. Adapting a brief dyadic intervention designed to target AUD to be delivered alongside COPE (COPE + B-FIT) is a promising way to bolster AUD outcomes and increase relationship functioning to promote recovery for Veteran and their families. The present study will test a modified version of B-FIT that is specifically designed to be delivered to Veterans with PTSD-AUD and their romantic partners. The goals of B-FIT are to: 1. increase reinforcement for AUD treatment engagement, 2. increase positive rewards from drinking reductions, and 3. decrease drinking cues by decreasing negative communication and increasing positive communication. This trial will recruit Veterans and their romantic partners (N=40 couples/80 individuals). This Stage 1a/1b trial will look at primary outcomes of feasibility and acceptability of the adapted B-FIT intervention, and secondary outcomes of PTSD symptoms, AUD symptoms, and psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Veterans and Significant Others:

* Any gender or sexual identity; any race or ethnicity
* Married, cohabiting for at least 6 months, or in a committed relationship for at least 6 months and both partners are willing to participate.
* The Veteran meets current or past-year DSM-5 diagnostic status for both PTSD (assessed via CAPS-5) and AUD (assessed via the Quick Structured Clinical Interview for DSM-5)

  * Concurrent substance use disorders are acceptable provided that alcohol is the Veteran's primary substance of choice
* Must demonstrate cognitive functioning sufficient to provide informed consent and participate accurately (=>26 on the Mini-Mental State Exam [MMSE])
* Participants taking psychotropic medications will be required to be maintained on a stable dose for at least 4 weeks before study initiation
* Not currently enrolled in couple therapy

Additional inclusion criteria for the Veteran patient:

* U.S. military Veteran
* Enrolled, or is willing to become enrolled, in VA healthcare
* Not attending trauma-focused therapy during the intervention period

Exclusion Criteria:

* History of moderate, severe, or unilateral violence in the relationship in the past year as measured by the CTS-2
* Either partner demonstrates a need for a higher level of care as assessed by the Quick Structured Clinical Interview for DSM-5 Disorders (QuickSCID)

  * i.e., history of or current psychotic or bipolar disorders, current severe drug use disorder, or concerns about alcohol withdrawal as demonstrated by a score >8 on the CIWA-Ar)
* Either partner reports current suicidal or homicidal ideation and intent or prior intent or attempt in the past 6 months as assessed by the CSSRS and PHQ-9 item 9
* The Veteran's SO cannot have substance use problems as indicated by a score < 8 on the AUDIT and QuickSCID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2027-03-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2031-02-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention to Participants (Customer Satisfaction Questionnaire) | at 12 weeks
  Veterans and Significant Others will report on their satisfaction with the adapted B-FIT intervention using the Customer Satisfaction Questionnaire (CSQ). Scores range from 1-4 and higher scores are indicative of greater satisfaction.
Feasibility of Intervention (Number of Sessions Attended) | Baseline to 12 weeks
  Feasibility of the adapted B-FIT intervention will be measured by number of sessions attended by each participant.

SECONDARY OUTCOMES:
Drinks per Drinking Day (Alcohol Timeline Followback (TLFB)) | Baseline to 12 weeks
  Change in drinks per drinking day, as measured by the Alcohol Timeline Followback (TLFB).
PTSD Symptoms (PTSD Checklist (PCL-5) | Baseline to 12 weeks
  Change in PTSD symptoms as measured by the PTSD Checklist (PCL-5). Scores range from 0-80 and higher scores are indicative of greater symptom severity.
Alcohol Problem Severity (Alcohol Use Disorders Identification Test (AUDIT)) | Baseline to 12 weeks
  Change in Alcohol problem severity as measured by the Alcohol Use Disorders Identification Test (AUDIT). Scores range from 0-40 with higher scores indicative of greater alcohol problem severity.
Relationship Satisfaction (Dyadic Adjustment Scales -7 (DAS-7)) | Baseline to 12 weeks
  Change in relationship satisfaction as measured by the brief Dyadic Adjustment Scales -7 (DAS-7). Scores range from 0-36, with higher scores indicating more positive relationship quality.
Quality of Life (Quality of Life Enjoyment and Satisfaction Scale (Q-LES-Q-SF)) | Baseline to 12 weeks
  Change in quality of life as measured by the Quality of Life Enjoyment and Satisfaction Scale (Q-LES-Q-SF). Scores range from 14-70 with higher scores indicating greater quality of life.
Interpersonal Functioning (Brief Inventory of Psychosocial Functioning (B-IPF)) | Baseline to 12 weeks
  Change in psychosocial functioning in relation to PTSD as measured by the Brief Inventory of Psychosocial Functioning (B-IPF). Scores range from 0-600 with higher scores indicating greater difficulty in psychosocial functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah T Giff, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No